CLINICAL TRIAL: NCT04526769
Title: Detecting SARS-CoV-2 Virus in Tears From Patients With COVID-19
Brief Title: Detecting SARS-CoV-2 in Tears
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: OVNS-2020-29066
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: COVID; COVID-19; Corona Virus Infection; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; Tear; Nasopharyngeal Swab
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Lacerations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Patients: All patients aged 18 years and above who present to Fairview/UMN ERs or ICUs with confirmed or suspect COVID-19 based on the attending physician's judgment will be included.
  Interventions: Diagnostic Test: Tear Collection

INTERVENTIONS:
Diagnostic Test: Tear Collection — A microcapillary tube will be placed at the corner of the eyelid so tears can be absorbed to the tube without causing any trauma. The tube will be placed in a transfer tube. Standard virus sampling swabs will be used to collect samples from the same patient's nasopharynx. RT-PCR will be run to determine virus yield in each sample.
  For the second part of the study, IHC staining will be done on the existing ocular tissue pathology slides to detect the expression of ACE2 and other cell surface and intracellular receptors. The investigators will use existing UMN ocular pathology lab and Lion's Eye Bank tissue samples. These are banked tissue samples that were collected and examined previously and then the remaining tissue samples were stored.

SUMMARY:
Purpose:

* To determine the presence of SARS-CoV-2 in tears
* To determine SARS-CoV-2 receptors in tear production system

DETAILED DESCRIPTION:
This is a prospective case series. NP swab and tear samples will be collected simultaneously from the confirmed or suspected COVID-19 patients. The samples will be transferred to the lab for SARS-CoV-2 testing. The presence of absence of SARS-CoV-2 will be compared in tears versus NP swabs.

The second part of the study is a histopathology examination series. Normal lacrimal gland and ocular surface tissue samples already stored at the UMN ocular pathology lab and Lion's Gift of Sight Eye Bank will be used for IHC staining for ACE2 and similar targets.

ELIGIBILITY:
Inclusion Criteria:

- Patients presenting at study sites with confirmed or suspected COVID-19

Exclusion Criteria:

* Pregnancy or nursing
* non-English speakers
* Those unable to read
* Those in other vulnerable study populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients meeting inclusion criteria who are willing to participate will be included until the total number of 30 participants is reached.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 Virus Detection in Tears | At day 1 of study participation
  Outcome is reported as the percent of tear samples that test either "positive", "negative", or "indeterminant" for SARS-CoV-2 Virus presence.
COVID-19 Virus Detection in Nasopharyngeal Swabs | At day 1 of study participation
  Outcome is reported as the percent of nasopharyngeal swab samples that test either "positive", "negative", or "indeterminant" for SARS-CoV-2 Virus presence.

SECONDARY OUTCOMES:
Expression of ACE2 in Lacrimal Gland Samples | At day 1 of study participation
  Pathology slides of lacrimal gland samples will be assessed for ACE2 expression and rated as having no expression (score=1), mild expression (score=2), or heavy expression (score=3). Outcome reported as the percent of lacrimal gland samples scored in each category (no expression, mild expression, or heavy expression).
Expression of ACE2 in Ocular Surface Samples | At day 1 of study participation
  Pathology slides of ocular surface samples will be assessed for ACE2 expression and rated as having no expression (score=1), mild expression (score=2), or heavy expression (score=3). Outcome reported as the percent of ocular surface samples scored in each category (no expression, mild expression, or heavy expression).

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Nazari, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided